CLINICAL TRIAL: NCT03953209
Title: Spironolactone for the Treatment of Melasma: a Prospective, Open-label Proof-of-concept and Dose-ranging Study
Brief Title: Spironolactone for the Treatment of Melasma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Conflict with funding
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00076765
Record Dates: First submitted 2019-04-18; First posted 2019-05-16 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Melasma
Keywords: spironolactone
MeSH Terms: conditions — Melanosis | interventions — Spironolactone; Tablets; Canrenoic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- spironolactone 50 mg (Experimental): Oral administration of spironolactone 50 mg once daily for 12 weeks
  Interventions: Drug: Spironolactone 50Mg Tablet
- spironolactone 100 mg (Experimental): Oral administration of spironolactone 100 mg once daily for 12 weeks
  Interventions: Drug: Spironolactone 100Mg Tablet
- spironolactone 200 mg (Experimental): Oral administration of spironolactone 200 mg once daily for 12 weeks
  Interventions: Drug: Spironolactone 200Mg

INTERVENTIONS:
Drug: Spironolactone 50Mg Tablet — Oral administration of one spironolactone 50 mg tablet once daily for 12 weeks
  Other Names: Aldactone
  Arms: spironolactone 50 mg
Drug: Spironolactone 100Mg Tablet — Oral administration of one spironolactone 100 mg tablet once daily for 12 weeks
  Other Names: Aldactone
  Arms: spironolactone 100 mg
Drug: Spironolactone 200Mg — Oral administration of two spironolactone 100 mg tablets once daily for 12 weeks
  Other Names: Aldactone
  Arms: spironolactone 200 mg

SUMMARY:
The purpose of this study is to prospectively gather data on the efficacy and tolerability of spironolactone to treat refractory melasma and to compare treatment response of randomized 50 mg, 100mg, and 200mg per day dosing.

DETAILED DESCRIPTION:
Melasma is a common, acquired condition of the skin characterized by symmetric reticulated hyperpigmented patches, most often of the central face and mandible.

An array of treatment modalities encompassing topical, oral, procedural, and combination therapies have been used to treat the disorder, with varying levels of immediate and long-term efficacy. Current treatment options are often unsuccessful in inducing complete disease remission. The tolerability of certain treatments is a valid concern, with adverse reactions such as irritation, peeling, burning, and post-inflammatory hyperpigmentation a common occurrence. Antiandrogens like spironolactone have been successfully used as adjunctive treatment for melasma. However, evidence for its off-label use for this purpose remains anecdotal. Clinical data regarding its efficacy and dosing are absent from the literature and are likely barriers to the drug's use in melasma. The high relapse rates and unfavorable side effect profiles of traditional treatment regimens underlie the need for an improved multimodal approach.

This prospective, randomized trial seeks to obtain information about the efficacy and tolerability of spironolactone to treat refractory melasma to guide future studies and clinical decision making. Participants will be randomized to one of the three dosage groups and take the study drug for 12 weeks. Outcomes will be assessed at baseline, week 6, week 12, and week 16. Subjects may opt to participate in a treatment extension period of up to 9 additional months, in which they will return to clinic monthly for outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have clinically diagnosed melasma, with an inadequate response to other treatment modalities, including but not limited to depigmenting agents, topical retinoids, topical steroids, peeling agents, laser and light therapies and combined topical creams.
2. Subject must be a female.
3. Subject must be 18-70 years of age.
4. Women of child-bearing potential must be on effective contraception. Acceptable methods of contraception include oral contraceptive pills (OCPs), hormonal or copper IUDs, contraceptive implants, contraceptive injections, birth control patches, vaginal rings, condom, sponge, diaphragm with spermicide, or prior surgical sterilization.
5. Subject must provide written informed consent prior to any study-related procedures being performed.
6. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

1. Subject is a pregnant or nursing female.
2. Subject has previously received spironolactone or another antiandrogenic treatment for melasma.
3. Subject is hyperkalemic, defined by a potassium level of greater than 5.1 mEq/liter.
4. Subjects with Addison's disease.
5. Subjects taking eplerenone or other potassium-sparing diuretics, lithium, cholestyramine, ACE inhibitors/angiotensin II antagonists/aldosterone blockers, or NSAIDS.
6. Subjects receiving potassium supplementation.
7. Subjects with history of renal disease or an eFGR < 30.
8. Subjects with acute or chronic liver failure.
9. Subject has an acute psychiatric condition that impairs ability to give consent or follow study protocols.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males will be excluded from this study due to the high incidence of gynecomastia and sexual dysfunction seen in spironolactone use at higher doses in men. The drug is not routinely used to treat dermatologic conditions in men due to its poor tolerability.
Enrollment: 0 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving clinical response | baseline and 12 weeks
  Clinical response defined as a 30% reduction in physician-assigned melanoma severity score on an anchored 100 mm visual analogue scale (VAS) with a minimum of 0 representing clear (better outcome) and a maximum of 100 representing very severe (worse outcome)

SECONDARY OUTCOMES:
Proportion of patients achieving clinical response | week 6, week 16, and optional treatment extension period visits lasting up to 1 yr
  Clinical response defined as a 30% reduction in physician-assigned melanoma severity score on an anchored 100 mm visual analogue scale (VAS) with a minimum of 0 representing clear (better outcome) and a maximum of 100 representing very severe (worse outcome)
Change in Dermatology Life Quality Index (DLQI) | baseline, week 6, week 12, week 16, and week 6, week 16, and optional treatment extension period visits lasting up to 1 yr
  Dermatology-specific quality of life questionnaire consisting of 10 items concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week. Each item is scored on a four point likert scale and the DLQI is calculated by summing the score of each question resulting in a minimum of 0 and a maximum of 30. The higher the score, the greater impairment of the patients QoL.
Tolerability of spironolactone as measured by incidence of treatment-related adverse events | baseline, week 6, week 12, week 16, and week 6, week 16, and optional treatment extension period visits lasting up to 1 yr
  Patient reported and physician observed
Comparing proportion of patients achieving clinical response between the three treatment arms: 50 mg, 100 mg, and 200 mg of spironolactone | week 6, week 12, week 16, and week 6, week 16, and optional treatment extension period visits lasting up to 1 yr
  Will estimate the difference between the proportions in the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elston, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No